CLINICAL TRIAL: NCT01653808
Title: In Vivo Evaluation of the Nipro Elisio™ Dialyzer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nipro Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nipro-Elisio 210H
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Kidney Disease
Keywords: CKD dialysis; hemodialysis; hemodiafiltration; Elisio dialyzer; efficacy; biocompatibility
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elisio-210H with HD (Experimental): hemodialysis patients treated with conventional hemodialysis (HD) modality using Elisio-210H dialyzer
  Interventions: Device: Elisio-210H; Procedure: conventional hemodialysis
- Elisio-210H with on line HDF (Active Comparator): hemodialysis patients treated with on line hemodiafiltration (HDF) modality using Elisio-210H dialyzer
  Interventions: Device: Elisio-210H; Procedure: on line hemodiafiltration

INTERVENTIONS:
Device: Elisio-210H — comparison of efficacy and biocompatibility of Elisio-210H dialyzer between conventional hemodialysis and on line hemodiafiltration
Procedure: conventional hemodialysis — comparison of conventional hemodialysis with on line hemodiafiltration using Elisio-210H dialyzer
  Arms: Elisio-210H with HD
Procedure: on line hemodiafiltration — comparison of on line hemodiafiltration with conventional hemodialysis using Elisio-210H dialyzer
  Arms: Elisio-210H with on line HDF

SUMMARY:
The purpose of this study is to compare the efficacy and biocompatibility of the Nipro Elisio 210H dialyzer between two dialysis modalities, conventional hemodialysis and on line hemodiafiltration.

DETAILED DESCRIPTION:
Hemodiafiltration, a convective-based therapy combining both diffusive and convective transports appears as the treatment modality of choice for hemodialysis patients. Indeed, this innovative technique offers an effective dialysis modality removing spectrum of uremic solutes with an optimized biocompatibility of the extracorporeal circuit obtained with use of ultrapure dialysis and sterile substitution fluids. However, such therapy can not be proposed in all dialysis centers due to major drawbacks of this technique over conventional hemodialysis, the complexity of the system and its increased costs. Alternatively, enhancement of convective transport may now be achieved by use of innovative dialyzers allowing more internal filtration. This is the case of ELISIO™-H dialyzers which possess fibers of a greater internal length which potentially allow more internal filtration. Aim of the present study was therefore to evaluate efficacy and biocompatibility of internal filtration-enhanced hemodialysis using this dialyzer compared to hemodiafiltration, over a four-month period.

ELIGIBILITY:
Inclusion Criteria:

* CKD dialysis patients on treatment with three times a week HD for more than three months
* with a stable anticoagulation scheme
* with haemoglobin level >10.5 g/dL
* with vascular access allowing a stable blood flow of 300 mL/min during treatment

Exclusion Criteria:

* patient already enrolled in another study
* pregnancy
* symptoms or signs of acute/chronic inflammatory or infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
pre-dialytic serum beta-2 microglobulin level | Month 1 (after one month)

SECONDARY OUTCOMES:
reduction rate of low molecular weight solutes (urea and creatinine) | Month 0, 1, 2, 3, 4
dialysis dose (urea KT/V) | Month 0, 1, 2, 3, 4
instantaneous clearance of low molecular weight solutes (urea and creatinine) | Month 0, 1, 2, 3, 4
inflammatory markers (CRP, fibrinogen, orosomucoide) | month 0, 1, 2, 3, 4
inflammatory marker (interkeukin 6) | month 0, 4
nutritional status (albumin, transthyretin, homocysteine) | Month 0, 1, 2, 3, 4
endothelial progenitor cells | Month 0, 1, 2, 3, 4
inflammatory mononuclear cell activation | Month 0, 1, 2, 3, 4
kappa and lambda light chains | Month 0, 4
oxidative stress parameters (superoxide anion, AOPPs, AGEs) | Month 0, 4
coagulation factors (TFPI, PAI-1, tPA, von willebrand factor and factor VIII) | Month 0, 4
apoptosis markers (soluble FAS and FAS ligand) | Month 0, 4
bone markers (bone PAL, Cross Laps, TRAP5b) | Month 0, 4

CONTACTS AND LOCATIONS:
Overall Officials: Bernard CANAUD, MD, Prof., Principal Investigator — University Hospital Center of Montpellier, France
Locations (1):
- University Hospital Center, Montpellier, France